CLINICAL TRIAL: NCT03266536
Title: Small Bowel Microbiota Characterization in Healthy Individuals Before and After Consumption of a Western Diet
Acronym: Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Colorado State University (Other); University of Minnesota (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-006388
Record Dates: First submitted 2016-10-26; First posted 2017-08-30 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Small Intestine Bacteria
Keywords: Gut microbiota
MeSH Terms: interventions — Diet, Western

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No western diet (No Intervention): Participants will undergo one-time testing for blood, urine, stool, and upper endoscopy with small bowel aspirates and biopsies. Participants will be finished with testing after the upper endoscopy is complete.
- Western diet (Experimental): Participants will undergo a first day of testing for blood, urine, stool, and upper endoscopy with small bowel aspirates and biopsies. Participants will then consume a Western diet for 7 days before a second day of identical testing (blood, urine, stool, and upper endoscopy with small bowel aspirates and biopsies).
  Interventions: Behavioral: Western diet

INTERVENTIONS:
Behavioral: Western diet — Western diet for 7 days: the meals in this Western diet will be provided by the Clinical Research and Trials Unit (CRTU) after participants meet with the nutrition staff (to discuss food preferences, how to obtain the meals). The meals will reflect a typical Western diet: a low fiber, high sugar diet with weight maintenance calories with < 10 grams fiber per day, and a typical US macronutrient calorie distribution of 50% carbs, 35% fat and 15% protein, with no alcohol. At least 50% of carbohydrates will be provided as simple sugars.
  Arms: Western diet

SUMMARY:
Does the small bowel microbiota in healthy individuals change after consumption of a Western diet?

DETAILED DESCRIPTION:
The gut microbiota is increasingly being implicated in disease. However, due to difficulty accessing the small bowel (i.e. requiring upper endoscopy) and the relative paucity of bacteria in this area (secondary to luminal flow and bactericidal bile acids/gastric acid), the small bowel microbiota is infrequently evaluated in any studies of this nature. The small bowel microbiota continues to remain an unexplored area of the gastrointestinal tract. Characterization of the microbial community and its function is the first step in determining how it potentially affects health and disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults between (and including) 18-65 years old.
* On a baseline healthy diet characterized by:

  * High fiber of ≥ 14 g/1000 calories/day
  * < 10% of daily calories from added sugar
  * At least 5 servings of fruit and vegetables per day
  * < or = 13% of daily calories from saturated fat

Exclusion Criteria:

* Patients who do not meet the above diet requirements.
* Known diagnosis of inflammatory bowel disease, microscopic colitis, celiac disease or other inflammatory conditions.
* Presence of abdominal symptoms based on baseline questionnaire.
* Commercial oral antibiotic or probiotic use within the past 4 weeks.
* Pregnancy or plans to become pregnant within the study time frame
* Vulnerable adults
* Any other disease(s), condition(s) or habit(s) that would interfere with completion of study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Transcriptional changes in gut microbiota present in stool. | Baseline, approximately three weeks.
  DNA extraction from stool samples will be done using standard assays.

CONTACTS AND LOCATIONS:
Overall Officials: Purna C Kashyap, M.B.B.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Principal investigator will protect the safety of subjects, the validity of data and the integrity of the research by assigning a study identification number to the subject. All information will be kept in a locked file cabinet and all data will be in a password protected computer database. All specimens will be stored in the principal investigator's freezer.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials